CLINICAL TRIAL: NCT02109523
Title: Improving Adherence to Medication After Coronary Artery Bypass Surgery (CABG) in Older Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir H Pakpour, Assistant Professor, Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 28/20/7200
Record Dates: First submitted 2014-04-01; First posted 2014-04-10 (Estimated); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Coronary Artery Bypass Grafting (CABG) Surgery
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Intervention (Experimental): Patients enrolled in the intervention arm will receive two educational sessions on the importance of medication and barriers to adherence
  Interventions: Behavioral: Motivational Interviewing (MI; Behavioral: volitional intervention
- Usual Care (Active Comparator): The usual care group received routine discharge counseling performed by the cardiologists and nurses.
  Interventions: Behavioral: Routine discharge counseling

INTERVENTIONS:
Behavioral: Motivational Interviewing (MI — Five weekly motivational and volitional session sessions and each last about 50 minutes. Five registered psychologists will moderated the session. All MI technique and planing intervention will be used.
  Other Names: facilitate behavior change
  Arms: Intervention
Behavioral: volitional intervention — Five weekly motivational and volitional session sessions and each last about 50 minutes. Five registered psychologists will moderated the session. All MI technique and planing intervention will be used.
  Other Names: Planning intervention
  Arms: Intervention
Behavioral: Routine discharge counseling
  Arms: Usual Care

SUMMARY:
Coronary artery bypass grafting (CABG) surgery is often performed in elderly patients, but non-adherence to post-CABG guideline medications is a common and serious clinical concern in this age group. A recent systematic review found that higher medication adherence significantly improved primary and secondary prevention of coronary artery disease outcomes in all the included studies. Another systematic review assessed studies published from 1999-2009 about motivational interviews, such as implementation intention, in relation to cardiovascular health. They found that motivational interview was an effective means of changing behavior, while offering promise in improving cardiovascular health status. The study is aimed to investigate effectiveness of long term volitional intervention in proving medication adherence in the CABG patient.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older
* Undergoing Elective/subacute multivessel CABG
* Able to give informed consent

Exclusion Criteria:

* Pregnant
* Already using Dosette boxes (or similar) to improve their medication adherence
* Currently enrolled in another clinical trial
* Unable to attend required follow-up visits
* Mini Mental Status Examination (MMSE) less than 20
* Significant dysphasia
* Concomitant surgery
* Myocardial infarction <48h of surgery
* Known platelet disease
* Allergic to aspirin
* Alcohol or narcotics abuse
* Geographically not available for follow up
* Ongoing bleeding
* Missing written consent
* Emergency surgery
* Severe kidney disease (creatinine clearance < 30 ml/min)
* Oxygen-dependent chronic obstructive pulmonary disease
* Active hepatitis
* Significant hepatic failure
* Prior peptic ulcer• Platelet count < 150 E9
* Patient has terminal condition and may not survive until 6-month follow-up
* Patient is a known participant in other RC studies
* The inability to read and write Persian/Farsi
* Participants who are not responsible for their own medication

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 288 (Actual)
Dates: Start 2014-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
changes in Patient-reported medication Adherence to four therapies (aspirin/antiplatelet; beta blocker; statin; ACE inhibitor) | changes from baseline , 6 Months, 12 months and 18 months after the intervention
Changes in Percent of Patients Adherent to four therapies (aspirin/antiplatelet; beta blocker; statin; ACE inhibitor) Via Refill Records | changes from baseline , 6 Months, 12 months and 18 months after the intervention

SECONDARY OUTCOMES:
Changes in psychological predictors of medication adherence (intention, perceived behavioral control and Self-monitoring) | changes from baseline, 6 Months, 12 months and 18 months follow-up
Changes in action planning | changes from baseline, 6 Months, 12 months and 18 months follow-up
  The number of planning strategies is used by the patients before, at baseline, six months, twelve months and eighteen months after the intervention
Changes in coping planning | changes from baseline, 6 Months, 12 months and 18 months follow-up
  The number of planning strategies is used by the patients before, at baseline, six months, twelve months and eighteen months after the intervention
Changes in quality of life | changes from baseline, 6 Months, 12 months and 18 months follow-up
Mortality rate and Myocardial Infarction | changes from baseline, 6 Months, 12 months and 18 months follow-up
Changes in Beliefs about Medications | changes from baseline, 6 Months, 12 months and 18 months follow-up
Changes in Illness Perceptions | changes from baseline, 6 Months, 12 months and 18 months follow-up
Changes in habit strength | changes from baseline, 6 Months, 12 months and 18 months follow-up
  Patient's habits on medications use before, at baseline, six months, twelve months and eighteen months after the intervention
Changes in total cholesterol | changes from baseline, 6 Months, 12 months and 18 months follow-up
Changes in blood pressure | changes from baseline, 6 Months, 12 months and 18 months follow-up
Changes in triglyceride | changes from baseline, 6 Months, 12 months and 18 months follow-up
Changes in high-density lipoproteins-cholesterol | changes from baseline, 6 Months, 12 months and 18 months follow-up
Changes in Low-density lipoproteins-cholesterol | changes from baseline, 6 Months, 12 months and 18 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Amir H Pakpour, PhD, Principal Investigator — Qazvin University Of Medical Sciences
Locations (13):
- Iran (13):
  - Golestan, Ahvāz
  - Mehr, Ahvāz
  - Booali Sina Hospital, Qazvin
  - Velayat Hospital, Qazvin
  - Kosar, Semnan
  - Shahid Madani, Tabriz
  - Firoozgar, Tehran
  - Imam Khomeini, Tehran
  - Rajaie, Tehran
  - Shariati, Tehran
  - Tehran Heart Center, Tehran
  - Khatam, Zahedan
  - Mousavi, Zanjan

REFERENCES:
- [Derived] Lin CY, Yaseri M, Pakpour AH, Malm D, Brostrom A, Fridlund B, Burri A, Webb TL. Can a Multifaceted Intervention Including Motivational Interviewing Improve Medication Adherence, Quality of Life, and Mortality Rates in Older Patients Undergoing Coronary Artery Bypass Surgery? A Multicenter, Randomized Controlled Trial with 18-Month Follow-Up. Drugs Aging. 2017 Feb;34(2):143-156. doi: 10.1007/s40266-016-0429-3. PMID 28004259